CLINICAL TRIAL: NCT00303615
Title: Androgen Therapy for Management of Estrogen/Progesterone Receptor Negative ER(-)PR(-) Metastatic Breast Cancer, Phase II Study
Brief Title: Androgen Therapy for Management of Estrogen/Progesterone Receptor Negative ER(-)PR(-) Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrural
Sponsor: Legacy Health System (Other)
Responsible Party: Nathalie Johnson, MD, Legacy Health System
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 200.3540
Record Dates: First submitted 2006-03-16; First posted 2006-03-17 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Metastatic Breast Cancer
Keywords: ER (-) and PR (-)
MeSH Terms: conditions — Breast Neoplasms | interventions — Fluoxymesterone; Anastrozole

INTERVENTIONS:
Drug: Fluoxymesterone 10 mg
Drug: Anastrozole 1 mg

SUMMARY:
This study is for patients with breast cancer that has spread to other tissues and organs. The purpose of this study is to identify patients who may respond favorably to certain types of hormonal therapy. Researchers will study your tumor, which was removed during your breast surgery. They will look for the presence or absence of Androgen (AR) receptors. These tests are for research purposes only. They will not affect the treatment of your breast cancer. The presence or absence of Androgen receptors on the tumor does not alter the therapy that is offered to patients. Recent evidence suggests that AR+ tumors are more likely to be destroyed when treated with androgen drugs. We will ask about 35 ER-/PR- breast cancer patients from Legacy Health System to be in this study. All tests and procedures are done as an outpatient in the doctor's office, a clinic, or at the hospital. The study drug that will be used in this trial is Androxy®, a synthetic androgen hormone. Androgens have been shown to inhibit the growth of some breast cancer cells. Arimidex is an aromatase inhibitor that will be used in conjunction with Androxy to inhibit the in vivo production of estrogen. It is hoped that the combination of these two drugs will inhibit the growth of your tumor and possibly cause it to shrink.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* ER Negative and PR Negative
* Progression of disease in the metastatic setting despite taxane or other chemotherapeutic therapies including Herceptin (patients on Herceptin may continue this therapy while on study)
* Maximized chemotherapy in the metastatic setting or patient experienced side effects contributing to decreased quality of life and elects to defer chemotherapy
* Evaluable disease by either:

  * CT Scan with or without contrast (lesions must be greater than 2 mm)
  * PET Scan, or Bone Scan, or Plain skeletal films
  * Chest wall or skin recurrence (digital photo to capture evaluable disease)
* Evaluable symptoms (pain, shortness of breath, fatigue, anorexia)
* Performance Status of 0, 1, or 2
* Bilateral mammogram performed within one year before registration

Exclusion Criteria:

* Uncontrolled hypercalcemia greater than 11
* Uncontrolled congestive heart failure greater than 2 NYHA class
* Central Nervous System metastasis
* Concomitant steroid use
* Performance Status of greater than 2
* Bilirubin greater than 5.5

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2005-06; Primary Completion 2007-06 (Estimated); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Time to disease progression

SECONDARY OUTCOMES:
Response of metastatic ER(-)PR(-) breast cancer to treatment with testosterone
Measure quality of life: improvement of fatigue in metastatic breast cancer patients
Measure degree of morbidity of treatment with testosterone in this setting

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Johnson, MD, Principal Investigator — Good Samaritan Foundation
Locations (1):
- Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon, United States